CLINICAL TRIAL: NCT00065442
Title: A Randomized, Double Blind, Placebo Controlled Phase 3 Trial of Immunotherapy With Autologous Antigen Presenting Cells Loading With PA2024 (Provenge(R), APC8015) in Men With Metastatic Androgen Independent Prostatic Adenocarcinoma
Brief Title: Provenge® (Sipuleucel-T) Active Cellular Immunotherapy Treatment of Metastatic Prostate Cancer After Failing Hormone Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dendreon (Industry)
Responsible Party: Liz Smith, Dendreon Corporation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D9902B; NCT00084760 (obsolete NCT alias)
Record Dates: First submitted 2003-07-23; First posted 2003-07-24 (Estimated); Results first posted 2010-09-06 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate; AIPC; androgen-independent; androgen independent; hormone insensitive; hormone-insensitive; PSA; prostatic adenocarcinoma; hormone-refractory; hormone refractory; HRPC; LHRH; immune therapy; immunotherapy; vaccine; dendritic cells; antigen-presenting cells; antigen presenting cells; cancer vaccine; therapeutic vaccine; therapeutic cancer vaccine; recombinant; biological; biopharmaceutical; biotechnology; biotech
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sipuleucel-T

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- APC-Placebo (Placebo Comparator)
  Interventions: Biological: APC-Placebo
- Sipuleucel-T (Active Comparator)
  Interventions: Biological: Sipuleucel-T

INTERVENTIONS:
Biological: Sipuleucel-T — Each dose of sipuleucel-T contains a minimum of 50 million autologous CD54+ cells activated with a PAP-GM-CSF. A course of therapy consists of 3 complete doses given at approximately 2-week intervals.
  Arms: Sipuleucel-T
Biological: APC-Placebo — Each dose of APC-Placebo contains approximately one-third of the quiescent APCs prepared from a single leukapheresis procedure. A course of therapy consists of 3 complete doses given at approximately 2-week intervals.
  Arms: APC-Placebo

SUMMARY:
Provenge is an investigational product designed to activate a man's own antigen presenting cells, a type of immune cell, so that they can detect prostate cancer cells and initiate an immune response against them.

Having completed Phase 1 and Phase 2 clinical trials, Provenge is now at the Phase 3 level. One important Phase 3 trial of Provenge has been completed; the current trial is also a Phase 3 study.

If you decide to participate and are eligible, you will be enrolled in the study and randomly assigned to receive either active product or placebo. There are two chances in three that you will receive Provenge. After receiving treatment, you will be monitored at regular intervals until the study endpoints are met. At the end of the trial, men who received placebo will have the opportunity to be treated with active product in another study.

DETAILED DESCRIPTION:
The trial is being conducted at multiple study centers throughout the United States. The trial is a double-blind, placebo-controlled trial. Participants must meet specific eligibility criteria. Study personnel will determine your eligibility in a telephone interview and through routine medical tests (physical exam, blood tests, imaging scans) done at a study center.

If you qualify for and decide to participate in the trial, you will have three product administrations over the course of one month.

ELIGIBILITY:
To qualify for this trial, you must have ALL of the following:

* Histologically documented adenocarcinoma of the prostate
* Cancer that has progressed while on adequate hormone therapy. This state of the disease is androgen independent prostate cancer (AIPC).
* Cancer that has spread outside the prostate (metastatic) to lymph nodes or bone. Please note that if your cancer has spread to organs (e.g., liver, lung, brain), you are not eligible for the study.
* The absence of or minimal current cancer-related pain

Please note that there are additional eligibility criteria. The study center will determine if you meet all of the criteria.

Study personnel will explain the trial in detail and answer any questions you may have if you do qualify for the study. You can then decide whether or not you wish to participate. If you do not qualify for the trial, study personnel will explain the reasons.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2003-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Schellhammer, MD, Study Chair — Devine Tidewater Urology
Locations (70):
- United States (64):
  - South Orange County Urological, Laguna Hills, California
  - LLUMC for Molecular Biology and Gene Therapy, Loma Linda, California
  - USC Keck School of Medicine, Los Angeles, California
  - UCLA, Los Angeles, California
  - Comprehensive Cancer Center, Palm Springs, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Group, San Diego, California
  - Sharp HealthCare, San Diego, California
  - UCSF Cancer Center, San Francisco, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Connecticut Urological Research at Grove Hill, New Britain, Connecticut
  - Helen F. Graham Cancer Center, Newark, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reid Army Medical Center, Washington D.C., District of Columbia
  - Miami Cancer Center, Miami, Florida
  - Urology Center of South Florida, Miami, Florida
  - Cancer Centers of Florida, Ocoee, Florida
  - Hematology/Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Georgia Urology, P.A., Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Midwest Prostate & Urology Health Center, Chicago, Illinois
  - Loyola University, Maywood, Illinois
  - Lutheran General Cancer Center, Park Ridge, Illinois
  - Indiana University, Indianapolis, Indiana
  - Chesapeake Urology Associates, Baltimore, Maryland
  - Myron I Murdock MD LLC, Greenbelt, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Clinic (Department of Urology), Burlington, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Associates in Urology, LLC, West Orange, New Jersey
  - Albany Regional Cancer Center, Albany, New York
  - The Urological Institute of Northeastern New York, Albany, New York
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - New York Medical College, Hawthorne, New York
  - Beth Israel Cancer Center, New York, New York
  - New York University, New York, New York
  - Clinical Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Staten Island Urological Research, Staten Island, New York
  - McKay Urology, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - EACRI, Portland, Oregon
  - Kaiser Permanente Medical Group, Portland, Oregon
  - Oregon Urology Specialists, Springfield, Oregon
  - Center for Urologic Care, Bryn Mawr, Pennsylvania
  - Jefferson Medical College, Philadelphia, Pennsylvania
  - Grand Strand Urology, Myrtle Beach, South Carolina
  - Mary Crowley, Dallas, Texas
  - Urology Associates of North Texas, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Urology of Virginia, PC, Norfolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - University of Wisconsin, Madison, Madison, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
  - St. Luke's Hospital Immunotherapy Program, Milwaukee, Wisconsin
- Canada (6):
  - Can-Med Medical Research, Inc., Victoria, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Urology CURC Scarborough, Scarborough Village, Ontario
  - Sunnybrook & Women's College HSC, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hospital Notre Dame du CHUM, Montreal, Quebec

REFERENCES:
- [Derived] Ju M, Fan J, Zou Y, Yu M, Jiang L, Wei Q, Bi J, Hu B, Guan Q, Song X, Dong M, Wang L, Yu L, Wang Y, Kang H, Xin W, Zhao L. Computational Recognition of a Regulatory T-cell-specific Signature With Potential Implications in Prognosis, Immunotherapy, and Therapeutic Resistance of Prostate Cancer. Front Immunol. 2022 Jun 23;13:807840. doi: 10.3389/fimmu.2022.807840. eCollection 2022. PMID 35812443
- [Derived] Small EJ, Higano CS, Kantoff PW, Whitmore JB, Frohlich MW, Petrylak DP. Time to disease-related pain and first opioid use in patients with metastatic castration-resistant prostate cancer treated with sipuleucel-T. Prostate Cancer Prostatic Dis. 2014 Sep;17(3):259-64. doi: 10.1038/pcan.2014.21. Epub 2014 Jun 24. PMID 24957547
- [Derived] Flanigan RC, Polcari AJ, Shore ND, Price TH, Sims RB, Maher JC, Whitmore JB, Corman JM. An analysis of leukapheresis and central venous catheter use in the randomized, placebo controlled, phase 3 IMPACT trial of Sipuleucel-T for metastatic castrate resistant prostate cancer. J Urol. 2013 Feb;189(2):521-6. doi: 10.1016/j.juro.2012.09.029. Epub 2012 Dec 14. PMID 23253957
- [Derived] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- See also: National Prostate Cancer Coalition — http://www.pcacoalition.org
- See also: USTOO International — http://www.ustoo.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized between August 2003 and November 2007 across 75 clinical trial sites.
Pre-assignment Details: Participants were screened for evaluation of subject eligibility and performance of baseline tests/procedures.
Groups:
- APC-Placebo: All subjects randomized to receive placebo. Approximately one-third of the quiescent APCs prepared from a single leukapheresis procedure. Three complete doses were given at approximately 2 week intervals.
- Sipuleucel-T: All subjects randomized to receive sipuleucel-T. Autologous peripheral blood mononuclear cells, including antigen presenting cells, that have been activated in vitro with a recombinant fusion protein, PAP-GM-CSF. Treatment consists of 3 doses administered approximately 2 weeks apart.
Period: Overall Study
Arm/Group | APC-Placebo | Sipuleucel-T
Started | 171 | 341
Completed | 46 | 121
Not Completed | 125 | 220
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 121 | 210
Not completed — Withdrawal by Subject | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | APC-Placebo | Sipuleucel-T | Total
Number analyzed (Participants) | 171 | 341 | 512
Age Continuous [Mean (Standard Deviation); unit: years] | 70.1 (9.0) | 71.1 (8.9) | 70.8 (8.9)
Age, Customized [Median (Full Range); unit: years] | 70 [40 to 89] | 72 [49 to 91] | 71 [40 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 171 | 341 | 512

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time from randomization until death due to any cause.
Time Frame: Event-driven timeframe. Final analysis at 331 events.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | APC-Placebo | Sipuleucel-T
Number analyzed (Participants) | 171 | 341
Months | 21.7 [17.7 to 23.8] | 25.8 [22.8 to 27.7]
Statistical Analysis 1: Comparison: APC-Placebo vs Sipuleucel-T; Test type: Superiority or Other; p = 0.032, Regression, Cox; Cox regression model with treatment, PSA (ln), and LDH (ln) as the independent variables, stratified by randomization strata; Hazard Ratio (HR) = 0.775, 95% CI 2-sided [0.614 to 0.979] — sipuleucel-T/placebo
Statistical Analysis 2: Comparison: APC-Placebo vs Sipuleucel-T; Test type: Superiority or Other; p = 0.023, Log Rank; Stratified by randomization strata; Hazard Ratio (HR) = 0.766, 95% CI 2-sided [0.608 to 0.965] — Cox regression model with treatment as the independent variable, stratified by randomization strata (sipuleucel-T/placebo)

2. Secondary Outcome: Time to Objective Disease Progression
Description: Measured by imaging studies; confirmed by independent imaging review
Time Frame: Analysis conducted at the time of overall survival analysis
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | APC-Placebo | Sipuleucel-T
Number analyzed (Participants) | 171 | 341
Weeks | 14.4 [11.7 to 15.0] | 14.6 [11.7 to 15.6]
Statistical Analysis 1: Comparison: APC-Placebo vs Sipuleucel-T; Test type: Superiority or Other; p = 0.628, Log Rank; Stratified by randomization strata; Hazard Ratio (HR) = 0.951, 95% CI 2-sided [0.773 to 1.169] — Cox regression model with treatment as the independent variable, stratified by randomization strata

ADVERSE EVENTS:
Time Frame: From randomization until time of overall survival analysis.
Description: Safety population: All subjects randomized to each arm who underwent at least one leukapheresis procedure. Not all randomized subjects underwent at least one leukapheresis procedure.
Arm/Group | APC-Placebo | Sipuleucel-T
Serious Adverse Events (participants affected / at risk) | 40/168 | 82/338
Other Adverse Events (participants affected / at risk) | 162/168 | 334/338
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APC-Placebo (N=168) | Sipuleucel-T (N=338)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 3
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 2
Cardiac tamponade (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
RECTAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 2
Catheter site haemorrhage (General disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Infusion related reaction (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 6
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Catheter bacteraemia (Infections and infestations) | 0 | 2
Catheter sepsis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 1 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Incision site infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 2 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Urinary tract infection Pseudomonal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Device malfunction (Injury, poisoning and procedural complications) | 0 | 1
Device occlusion (Injury, poisoning and procedural complications) | 1 | 1
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Brain scan abnormal (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain mass (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 6
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 2 | 4
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Bladder obstruction (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 2 | 2
Hydronephrosis (Renal and urinary disorders) | 2 | 1
Obstructive uropathy (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 4 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Reexpansion pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Pallor (Vascular disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | APC-Placebo (N=168) | Sipuleucel-T (N=338)
Anaemia (Blood and lymphatic system disorders) | 21 | 50
Constipation (Gastrointestinal disorders) | 24 | 45
Diarrhoea (Gastrointestinal disorders) | 17 | 36
Nausea (Gastrointestinal disorders) | 35 | 95
Vomiting (Gastrointestinal disorders) | 20 | 60
Asthenia (General disorders) | 13 | 37
Chills (General disorders) | 21 | 183
Fatigue (General disorders) | 64 | 132
Influenza like illness (General disorders) | 6 | 33
Oedema peripheral (General disorders) | 16 | 32
Pain (General disorders) | 12 | 44
Pyrexia (General disorders) | 23 | 99
Upper respiratory tract infection (Infections and infestations) | 9 | 15
Urinary tract infection (Infections and infestations) | 12 | 22
Citrate toxicity (Injury, poisoning and procedural complications) | 34 | 68
Contusion (Injury, poisoning and procedural complications) | 9 | 9
Weight decreased (Investigations) | 18 | 20
Anorexia (Metabolism and nutrition disorders) | 27 | 24
Decreased appetite (Metabolism and nutrition disorders) | 11 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 | 70
Back pain (Musculoskeletal and connective tissue disorders) | 61 | 116
Bone pain (Musculoskeletal and connective tissue disorders) | 18 | 32
Flank pain (Musculoskeletal and connective tissue disorders) | 10 | 9
Muscles spasms (Musculoskeletal and connective tissue disorders) | 9 | 24
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 19 | 33
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20 | 44
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 33
Neck pain (Musculoskeletal and connective tissue disorders) | 7 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 | 49
Dizziness (Nervous system disorders) | 16 | 49
Headache (Nervous system disorders) | 8 | 54
Hypoaesthesia (Nervous system disorders) | 5 | 18
Paraesthesia (Nervous system disorders) | 26 | 45
Paraesthesia oral (Nervous system disorders) | 21 | 41
Anxiety (Psychiatric disorders) | 14 | 13
Depression (Psychiatric disorders) | 11 | 8
Insomnia (Psychiatric disorders) | 12 | 24
Haematuria (Renal and urinary disorders) | 9 | 31
Hydronephrosis (Renal and urinary disorders) | 12 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 28
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 18
Rash (Skin and subcutaneous tissue disorders) | 9 | 16
Hypertension (Vascular disorders) | 5 | 25
Hypotension (Vascular disorders) | 9 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A provision provides for sponsor review up to 45 days with the right to request modification based on disclosure of confidential information; extendable by 60 days to file a patent application.